CLINICAL TRIAL: NCT06960174
Title: Virtual Renality: Assessing the Impact of Virtual Reality on Preoperative Planning in Renal Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Hille Torenvlied, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL-009626
Record Dates: First submitted 2025-04-18; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer)
Keywords: Renal Cell Carcinoma; Partial nephrectomy; Radical nephrectomy; Preoperative planning; 3D virtual model; Virtual Reality
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative planning based on CT (No Intervention): For the control group the preoperative planning will be according to the current standard of care using only the CT scan.
- Preoperative planning based on CT + VR (Experimental): For the intervention group, the urologist will review a 3D virtual model of the renal anatomy in addition to the CT scan during preoperative planning
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — If the participant is assigned to the intervention group a 3D virtual model will be constructed. For the intervention group the CT + VR will be reviewed during preoperative planning.
  Arms: Preoperative planning based on CT + VR

SUMMARY:
Rationale:

Preoperative planning for both partial and radical nephrectomies using conventional CT imaging can be challenging due to complex renal anatomy and vascularization. 3D models in virtual reality (VR) may enhance anatomical understanding and improve preoperative planning. This study aims to prospectively evaluate the clinical impact of the use of 3D models in VR in the preoperative planning of partial and radical nephrectomies.

Objective:

The primary objective is to assess the impact of VR on preoperative planning and thereby on the agreement between the preoperative plan and the performed surgery in renal surgery (both partial and radical nephrectomies). The secondary objectives focus on the urologist's understanding of the anatomy and how the intraoperative and postoperative outcomes are influenced by the use of VR in the preoperative planning.

Study design:

The Virtual Renality study is a single-center randomized clinical trial conducted at the St. Antonius Hospital in Nieuwegein.

Study population:

The study population will consist of adult patients (18+) with a suspected RCC who are indicated for (partial) nephrectomy at St. Antonius Hospital Nieuwegein.

Intervention:

For the intervention group, the urologist will review a 3D virtual model of the renal anatomy in addition to the original CT scan during preoperative planning. For the control group, only the CT scan will be used for preoperative planning, according to the current standard of care.

Main study parameters/endpoints:

The primary study endpoint is the surgical concordance score, which describes the concordance between the actual performed surgery and the preoperatively determined surgical plan.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness:

Participation in this study will not require any additional physical examinations, blood samples, hospital visits, or questionnaires beyond standard clinical care. The only difference for participants in the intervention group is that a 3D model will be created from the existing CT scan and reviewed in VR during preoperative planning by the urologist.

DETAILED DESCRIPTION:
The Virtual Renality study is a single-center randomized clinical trial conducted at the St. Antonius Hospital in Nieuwegein. For the intervention group, the urologist will review a 3D virtual model of the renal anatomy in addition to the original CT scan during preoperative planning, whereas for the control group, only the CT scan will be used for preoperative planning, according to the current standard of care. The flowchart in Figure 1 provides an overview of the study design. The steps covered in the flowchart and the collection of parameters will be further explained later in this protocol. The study is single-blinded, as the 3D virtual model during preoperative planning is the assessed intervention. Participants will be randomly assigned to either the control group or the intervention group to eliminate selection bias and achieve comparability between the two groups. The urologists who perform (partial) nephrectomies at the St. Antonius Hospital will participate in the study. A total of 72 patients suspected of having a renal tumor and indicated for (partial) nephrectomy will be included. The inclusion period for the study will take approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* 18+
* Suspected RCC and candidate for (partial) nephrectomy
* Signed informed consent

Exclusion Criteria:

* Patients who are not approved to undergo surgery (due to comorbidities or their overall health condition)
* Patients who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Concordance score between actual performed surgery and surgical plan | during preoperative planning (approximately 3 days before surgery) and immediately after surgery
  To assess whether the surgery is performed according to the preoperative plan, a questionnaire regarding the expected surgical steps will be completed during the preoperative planning. Postoperatively, the data will be collected from the surgical notes. The postoperative data will be compared with the preoperatively filled questionnaire and this will result in a concordance score between the actual performed surgery and the preoperatively determined surgical plan. This score of concordance will be the primary study endpoint

SECONDARY OUTCOMES:
Intra-operative parameters: method of clamping | Perioperative
  Method of clamping (main renal artery / multiple arteries / no clamping / selective clamping)
Intraoperative parameters: blood loss | Perioperative
  blood loss (value in ml)
Intraoperative parameters: clamping time | Perioperative
  clamping time (value in mm:ss)
Intraoperative parameters: opening of collecting system | Perioperative
  opening of collecting system (yes/no)
Intraoperative parameters: duration of surgery | Perioperative
  duration of surgery (value in minutes)
Post-operative parameters: renal function | Up to 1 month post-surgery
  Renal function (Creatinine level before surgery, 1 day post-surgery and 4 weeks post-surgery )
Post-operative parameters: 30-day post-surgery complications | 30 days post-surgery
  30-day post-surgery complications ( Clavien Dindo score (Grade I / Grade II / Grade IIIa / Grade IIIb / Grade IVa / Grade IVb / Grade V) )
Post-operative parameters: hospital stay | 30-days post-surgery
  hospital stay (days)
Post-operative parameters: readmission (within 30 days) | 30-days post-surgery
  readmission (within 30 days) (yes/no)
Post-operative parameters: clean resection margin | 30-days post-surgery
  clean resection margin (yes/no)
Post-operative parameters: | 30-days post-surgery
  pathological TNM (TxNxMx)
Understanding of anatomy - renal arteries | during preoperative planning (approximately 3 days before surgery) and immediately after surgery
  Understanding of renal arteries (Very poor / Poor / Moderate / Good / Excellent)
Understanding of anatomy - renal veins | during preoperative planning (approximately 3 days before surgery) and immediately after surgery
  Understanding of renal veins (Very poor / Poor / Moderate / Good / Excellent)
Understanding of anatomy - collecting system | during preoperative planning (approximately 3 days before surgery) and immediately after surgery
  Understanding of collecting system (Very poor / Poor / Moderate / Good / Excellent)
Understanding of anatomy - tumor | during preoperative planning (approximately 3 days before surgery) and immediately after surgery
  Understanding of tumor anatomy (Very poor / Poor / Moderate / Good / Excellent)
Understanding of anatomy - general anatomy | during preoperative planning (approximately 3 days before surgery)
  Confidence in understanding of general anatomy (Strongly disagree / Disagree / Neutral / Agree / Strongly agree)

OTHER OUTCOMES:
Demographic data - age | before surgery
  Age (Years (at time of surgery) )
Demographic data - gender | before surgery
  Gender (Male / Female )
Medical data - BMI | before surgery
  BMI (Kg/m2)
Medical data - ASA-score | before surgery
  ASA-score ( I / II / III / IV / V)
Medical data - history of smoking | before surgery
  History of smoking (Packyears (or yes/no) )
Medical data - comorbidities | before surgery
  Comorbidities (Charlson comorbidity index, 0-37))
Medical data - radiological TNM | before surgery
  Radiological TNM classification (TxNxMx )
Medical data - RENAL | before surgery
  RENAL score (4-12 a/p/h)
Medical data - tumor side | before surgery
  Side of tumor(Left/right)
Medical data - tumor size | before surgery
  Size of tumor (mm)
Medical data - CT type | before surgery
  Type of CT (Contrast enhanced (which phases)/photon counting)
Medical data - surgeon | before surgery
  Surgeon (Name / number )